CLINICAL TRIAL: NCT04062318
Title: The Causal Role of Neocortical Beta Events in Human Sensory Perception
Brief Title: Beta Events and Sensory Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1902002327; P20GM103645 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Beta Rhythm; Tactile Perception
Keywords: somatosensory; tactile; perception; electroencephalography; transcranial magnetic stimulation; beta rhythm

STUDY DESIGN:
Intervention Model Description: All participants will complete an initial MRI. MRIs are subsequently used for TMS neuronavigation (region of interest targeting). There is no intervention applied during the MRI session.
  In two subsequent concurrent TMS-EEG sessions, all participants will receive active TMS while carrying out a tactile detection task. During one of the two TMS-EEG sessions, TMS will be applied over primary somatosensory cortex. During the other TMS-EEG session, TMS will be applied over a control brain region.
  The order of somatosensory vs. non-somatosensory TMS targeting will be counterbalanced across participants.
Who Masked: Participant
Masking Description: Participants will be unaware of the order in which they receive TMS interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tactile detection task with online TMS-EEG (Experimental): Participants receive perceptual threshold-level tactile stimuli to the third digit of the right hand and report detection or non-detection. EEG is recorded and TMS is applied over somatosensory cortex during the tactile detection task.
  Interventions: Device: Online active TMS
- Tactile detection task with online control TMS-EEG (Active Comparator): Participants receive perceptual threshold-level tactile stimuli to the third digit of the right hand and report detection or non-detection. EEG is recorded and TMS is applied over a control brain region during the tactile detection task. This control condition is intended to mimic the peripheral (e.g. cranial/facial muscle and/or nerve activation, auditory evoked response), but not biological effects of TMS specifically related to somatosensory perception.
  Interventions: Device: Online active TMS

INTERVENTIONS:
Device: Online active TMS — One single pulse or triple pulse train (3 pulses, 20ms inter-pulse interval) of TMS will be delivered per trial (at least 5 seconds apart) "online", or during the tactile detection task, at less than or equal to 80% active motor threshold.

SUMMARY:
Low-frequency brain rhythms in the alpha (8-14Hz) and beta (15-29Hz) bands are strong predictors of perception and functional performance in a range of tasks, and are disrupted in several disease states. The purpose of this study is to investigate a direct causal relationship between low-frequency brain rhythms and sensory perception, and to optimize commonly used TMS paradigms to impact sensory processing and perception in a similar manner as endogenous rhythms. To do so, this study combines human magnetic resonance imaging (MRI), electroencephalography (EEG), non-invasive brain stimulation (transcranial magnetic stimulation; TMS), and biophysically principled computational neural modeling.

DETAILED DESCRIPTION:
Prior studies have shown that high power low-frequency brain rhythms in the alpha (8-14) and beta (15-29 Hz) bands in primary somatosensory cortex (SI) are associated with a decreased probability of perceiving tactile stimuli at perceptual threshold, and can be modulated with attention. Furthermore, high power beta activity in SI emerges as brief "events" (<150ms) in un-averaged data, the rate and timing of which underlie the attentional and perceptual effects associated with high beta power.

In this study, human electroencephalography (EEG) and a non-painful tactile detection task are used to assess if and how the rate and timing of ongoing rhythmic events in the alpha/beta bands prior to a tactile stimulus causally impact touch perception, and how this relates to attention. A custom TMS protocol that is hypothesized to mimic endogenous beta-frequency event patterns is used to test whether TMS can impact perception in a similar manner. Finally, computational neural modeling designed to simulate macro-scale EEG signals is used to aid in the interpretation of potential neural circuit mechanisms underlying features of acquired EEG data.

The TMS-EEG components of this study will use a within-subjects crossover design. In initial study sessions, participants will have an MRI. In subsequent study sessions, participants will complete a tactile detection task while EEG data is recorded concurrent with online active or sham TMS. Analyses will focus on comparing detection probabilities of tactile stimuli presented at perceptual threshold and tactile evoked response potential waveforms between trials in which TMS pulses or endogenous beta events occur with similar timing and intensity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent/assent
* Age: 18-65 years
* English fluency: participants must be able to understand screening questionnaires and task instructions spoken/written in English.
* Right handed: to reduce heterogeneity related to hand dominance, since our task involves touch perception on the hand, and examination of neural correlates in lateralized brain regions.

Exclusion Criteria:

* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy
* Any progressive (e.g., neurodegenerative) neurological disorder
* Chronic medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* Metal implants (excluding dental fillings)
* Pacemaker
* Implanted medication pump or cochlear implant
* Vagal nerve stimulator
* Deep brain stimulator
* TENS unit (unless removed completely for the study)
* Ventriculo-peritoneal shunt
* Signs of increased intracranial pressure
* Intracranial lesion
* History of head injury resulting in prolonged loss of consciousness
* Pregnancy
* Participants who have received prior TMS for medical treatment purposes.
* Intellectual Disability or autism spectrum disorder (ASD)
* Active psychosis, diagnosis of unipolar depression or bipolar disorder, active severe substance use disorders (within the last month), or active suicidal intent or ideations.
* Conditions that may result in the inability to effectively carry out the tactile detection task, including loss of feeling, neuropathy or nerve damage in the hands or feet, chronic pain or fibromyalgia, and pain due to cancer, infection or arthritis.
* If the participant is actively taking any of the medications that increase risk from TMS as indicated below, of if they have ingested any alcohol or any other drugs of abuse (see https://www.drugabuse.gov/drugs-abuse) on the day of the study session (prior to the session).

Contraindicated medications:

alcohol Amitriptyline Amphetamines ampicillin Anticholinergics Antihistamines aripiprazole BCNU **bupropion** cephalosporins chlorambucil chloroquine Chlorpromazine citalopram Clozapine Cocaine cyclosporine cytosine arabinoside Doxepine duloxetine fluoxetine fluphenazine fluvoxamine Foscarnet gamma-hydroxybutyrate (GHB) Ganciclovir haloperidol imipenem Imipramine isoniazid ketamine levofloxacin Lithium Maprotiline MDMA (ecstasy) mefloquine methotrexate metronidazole mianserin mirtazapine Nortriptyline olanzapine paroxetine penicillin phencyclidine (PCP, angel's dust) pimozide quetiapine reboxetine risperidone Ritonavir **Sertraline** Sympathomimetic theophylline venlafaxine vincristine ziprasidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Threshold-level tactile detection | Measures of tactile detection are collected during the tactile detection task, which is assessed on each study visit (with the exception of an MRI-only visit) throughout the course of study completion, an average of 6-12 months.
  Participants receive one tactile stimulus per trial and report detection or non-detection using a button press. Stimuli are delivered at one of three intensities: perceptual threshold-level (70% of trials), suprathreshold-level (always perceived, 10% of trials) or null stimuli (no stimulus, 20% of trials).
EEG tactile evoked response potential (ERP) | EEG measures are collected during the tactile detection task, which is assessed on each study visit (with the exception of an MRI-only visit) throughout the course of study completion, an average of 6-12 months.
  Participants receive one tactile stimulus per trial concurrent with EEG recording. The EEG-measured ERP immediately following each tactile stimulus is assessed and compared across conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R Jones, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Carney Institute for Brain Science Human Testing Space (HuTS), Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones SR, Kerr CE, Wan Q, Pritchett DL, Hamalainen M, Moore CI. Cued spatial attention drives functionally relevant modulation of the mu rhythm in primary somatosensory cortex. J Neurosci. 2010 Oct 13;30(41):13760-5. doi: 10.1523/JNEUROSCI.2969-10.2010. PMID 20943916
- [Background] Sherman MA, Lee S, Law R, Haegens S, Thorn CA, Hamalainen MS, Moore CI, Jones SR. Neural mechanisms of transient neocortical beta rhythms: Converging evidence from humans, computational modeling, monkeys, and mice. Proc Natl Acad Sci U S A. 2016 Aug 16;113(33):E4885-94. doi: 10.1073/pnas.1604135113. Epub 2016 Jul 28. PMID 27469163
- [Background] Shin H, Law R, Tsutsui S, Moore CI, Jones SR. The rate of transient beta frequency events predicts behavior across tasks and species. Elife. 2017 Nov 6;6:e29086. doi: 10.7554/eLife.29086. PMID 29106374
- [Background] Jones SR, Pritchett DL, Stufflebeam SM, Hamalainen M, Moore CI. Neural correlates of tactile detection: a combined magnetoencephalography and biophysically based computational modeling study. J Neurosci. 2007 Oct 3;27(40):10751-64. doi: 10.1523/JNEUROSCI.0482-07.2007. PMID 17913909
- [Background] Jones SR, Pritchett DL, Sikora MA, Stufflebeam SM, Hamalainen M, Moore CI. Quantitative analysis and biophysically realistic neural modeling of the MEG mu rhythm: rhythmogenesis and modulation of sensory-evoked responses. J Neurophysiol. 2009 Dec;102(6):3554-72. doi: 10.1152/jn.00535.2009. Epub 2009 Oct 7. PMID 19812290